CLINICAL TRIAL: NCT02383394
Title: Factors Associated With Second-Trimester Pregnancy Loss in Women With Normal Uterine Anatomy Undergoing In Vitro Fertilization
Brief Title: Factors Associated With Pregnancy Loss in IVF Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Other Study IDs: 131
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Invitro Fertilization
Keywords: second trimesteric pregnancy loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- aborted women: women who got pregnant and have 2nd trimesteric abortion, follow up antenatal care by ultrasound and clinical monitoring
  Interventions: Other: follow up antenatal care
- continued women: women who got pregnant and completed her pregnancy follow up antenatal care by ultrasound and clinical monitoring
  Interventions: Other: follow up antenatal care

INTERVENTIONS:
Other: follow up antenatal care — ultrasound follow up of pregnancy

SUMMARY:
Maternal and clinical characteristics associated with spontaneous second-trimester pregnancy loss (between 12 1/7 and 23 6/7 weeks of gestation) will be assessed.

DETAILED DESCRIPTION:
Maternal characteristics as age , parity, body mass index, previous abortion,previous failed IVF cycles, weight gain during pregnancy, physical activity, sexual relation and frequency, adherence to treatment, residency, medical history,surgical pelvic history, fever during pregnancy.

Clinical characteristics as multiple pregnancy, site of implantation, day of transfer, serum HCG day 14.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 21-44 years with ongoing in vitro fertilization pregnancy (at least one fetus with fetal heart tones at 12 weeks of gestation)

Exclusion Criteria:

* abnormal uterine cavity induced abortion for medical problem

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged 21-44 years with ongoing in vitro fertilization pregnancy (at least one fetus with fetal heart tones at 12 weeks of gestation)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2017-05 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
second trimester abortion | between 12 1/7 and 23 6/7 weeks of gestation)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Ahmed Maged, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes